CLINICAL TRIAL: NCT03023514
Title: Lipoic Acid Supplementation in IVF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized
Other Study IDs: ALA_ImplRate
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Women Infertility
Keywords: Oocyte donation; IVF; Lipoic acid; Implantation rate; Endometrial receptivity
MeSH Terms: interventions — Thioctic Acid

ARMS (2):
- ALA + P (Experimental): Oral alpha-lipoic acid + vaginal Progesterone
  Interventions: Dietary Supplement: Oral Lipoic acid; Drug: Vaginal Progesterone
- P (Active Comparator): vaginal Progesterone
  Interventions: Drug: Vaginal Progesterone

INTERVENTIONS:
Dietary Supplement: Oral Lipoic acid — 300 mg ALA x2 (1pill orally/12h) to the recipient from the day of the donors pick up until 8 week of pregnancy
  Arms: ALA + P
Drug: Vaginal Progesterone — 200 mg Vaginal Progesterone (1 vaginal capsule/24h) from the day of the donors pick up until 8 week of pregnancy

SUMMARY:
Alpha-Lipoic Acid (ALA) is a natural molecule that can make a significant contribution to the success of embryo implantation phase, because it exerts, directly or indirectly, an immunomodulatory activity. ALA has the ability to regenerate antioxidants molecules that facilitate embryo implantation, and to stimulate the production of local mediators useful for implantation. This study is a prospective clinical trial and aims to evaluate the reproductive outcomes of Italian couples following oocyte donation fresh cycles when receiving per os tablets of lipoic acid. Indeed, the control group had only the standard treatment (vaginal progesterone), whereas the study group, in addition to that, received ALA (300 mg, 2 times per day) by oral route, from the day of donors oocyte pick up until the pregnancy test. If the childbearing occurred, treatment continued until the 8th week of pregnancy. Primary outcome of the study is the implantation rate while the positive hCG rate, the clinical pregnancy rate, the miscarriage rate and the live-birth rate are secondary outcomes .

ELIGIBILITY:
Inclusion Criteria:

Donors:

* Proof of fertility;
* ⩽32 years old
* BMI <30 kg/m2
* Regular menstrual cycles of 25-33 days
* Two normal ovaries based on transvaginal scan findings.

Recipients:

* Women with infertility problems
* ⩽50 years old,
* BMI <34 kg/m2

Exclusion Criteria:

Donors:

* Polycystic ovaries
* Endometriosis
* Gynaecological or medical disorders.

Recipients:

* Endocrinologic problems
* Medication for chronic illness
* Azoospermic partner that require TESE
* Sperm donation cycles

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of implants per cycle | Within 7 weeks after blastocystis transfer
  Implantation rate is defined as the percentage of transferred embryos that develop at least to the stage of fetal heart activity documented by pregnancy ultrasound.

SECONDARY OUTCOMES:
Number of biochemical pregnancies per group | Within 7 weeks after blastocystis transfer
  Positive β-human chorionic gonadotropin (hCG) test
Number of clinical pregnancies per group | 7 weeks of gestation
  A positive β-hCG test and a fetal heart beat seen by ultrasound at 7 weeks of gestation was defined as a clinical pregnancy, otherwise it was considered a biochemical pregnancy.
Number of live birth per group | At delivery
Number of miscarriage per group | Within 22 weeks of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Iakentro Advanced Medical Centre, IVF Unit, Thessaloniki, Greece

REFERENCES:
- [Background] Monastra G, De Grazia S, Cilaker Micili S, Goker A, Unfer V. Immunomodulatory activities of alpha lipoic acid with a special focus on its efficacy in preventing miscarriage. Expert Opin Drug Deliv. 2016 Dec;13(12):1695-1708. doi: 10.1080/17425247.2016.1200556. Epub 2016 Jun 24. PMID 27292272
- [Background] Cha J, Sun X, Dey SK. Mechanisms of implantation: strategies for successful pregnancy. Nat Med. 2012 Dec;18(12):1754-67. doi: 10.1038/nm.3012. PMID 23223073